CLINICAL TRIAL: NCT05298228
Title: Dose Finding Study of Remimazolam for Laryngeal Mask Airway Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4-2021-1706
Record Dates: First submitted 2022-03-06; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Orthopedic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remimazolam (Experimental): A bolus dose of remimazolam is administered to facilitate LMA insertion
  Interventions: Drug: Remimazolam bolus does administration

INTERVENTIONS:
Drug: Remimazolam bolus does administration — The beginning dose of remimazolam is 0.3 mg/kg, and when LMA insertion is successful, the dose will be decreased by 0.05 mg/kg in the next patient. When LMA insertion is unsuccessful (failed), the dose will be increased by 0.05 mg/kg in the next patient.

SUMMARY:
Laryngeal mask airways (LMA) are widely used in patients receiving general anesthesia and are known to have the following advantages over the endotracheal tube: lower incidence of postoperative sore throat, lower incidence of cough during emergence, and lower incidence of postoperative vomiting. Although LMAs can be inserted without the use of muscle relaxants, a sufficient depth of anesthesia is necessary for placement. Remimazolam is a newer anesthetic that is ultra-short acting with a rapid onset and short context-sensitive half-life allowing for fast recovery. However, the dose of remimazolam needed for LMA insertion without muscle relaxants is not well known. This dose-finding study aims to find the ED50 and ED95 of a single bolus dose of remimazolam for LMA insertion without muscle relaxants in adult patients.

This is an interventional study done in a single group using the Dixon's up-and-down method which requires at least six success/failure pairs in the same direction. The primary endpoint of this study is to investigate the dose of remimazolam associated with 50% (ED50) and 95% (ED95) probability for adequate depth of anesthesia for LMA insertion without muscle relaxants. The beginning dose of remimazolam is 0.3 mg/kg, and when LMA insertion is successful, the dose will be decreased by 0.05 mg/kg in the next patient. When LMA insertion is unsuccessful (failed), the dose will be increased by 0.05 mg/kg in the next patient. Successful LMA insertion is defined as symmetrical chest wall movement and square-wave capnographic traces observed with manual ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19~65 year
* ASA class I~III
* Patients scheduled for orthopedic surgery under general anesthesia and eligible for LMA use.

Exclusion Criteria:

* Patient refusal
* Patients unable to read consent form
* Anticipated difficult mask ventilation
* Active URI or uncontrolled asthma
* Pneumonia
* Risk of aspiration such as GERD
* History of allergies to benzodiazepines
* Decreased liver or kidney function
* Pregnant or breastfeeding patients
* BMI > 30kg/m2
* History of substance abuse/addiction

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-07-26 (Estimated); Study Completion 2023-07-27 (Estimated)

PRIMARY OUTCOMES:
Dose of remimazolam associated with 50% (ED50) probability for adequate depth of anesthesia for LMA insertion without muscle relaxants. | During procedure (Immediately after LMA insertion attempt)
  The primary outcome of this study will be determined based on the data of "success" or "failure" of LMA insertion at predetermined doses of remimazolam. Successful LMA insertion is defined as symmetrical chest wall movement and square-wave capnographic traces observed with manual ventilation which will be assessed immediately after LMA insertion attempt.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho E, Roh YH, Moon J, Kim Y, Shin S. Effective bolus dose of remimazolam for i-gel(R) insertion in nonparalyzed patients: a dose-finding study. Can J Anaesth. 2024 Sep;71(9):1251-1260. doi: 10.1007/s12630-024-02762-w. Epub 2024 Apr 26. PMID 38671251